CLINICAL TRIAL: NCT07371884
Title: The Effect of Dramatic Play on Bullying Behaviors in Preschool Children
Brief Title: Dramatic Play and Bullying Behaviors in Preschool Children
Acronym: DRAMA-BULLY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Devran ATALAY ÖZKILIÇ, Principal Investigator, Ataturk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ATATURKU-HF-DAÖ-01
Record Dates: First submitted 2026-01-07; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Bullying Behavior; Aggressive Behavior
Keywords: peer bullying; dramatic play; preschool children
MeSH Terms: conditions — Aggression

STUDY DESIGN:
Intervention Model Description: All students will be accepted.
Masking Description: Data collection tools will be collected by an interviewer independent of the research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dramatic play application (Experimental): In this group, dramatic play activities aimed at reducing bullying behaviors will be implemented for preschool children.
  Interventions: Behavioral: dramatic play intervention

INTERVENTIONS:
Behavioral: dramatic play intervention — A dramatic play program will be implemented to reduce bullying behaviors in preschool children. The intervention will consist of structured dramatic play activities aimed at developing social interaction, empathy, and problem-solving skills, and will be implemented over a period of 10 weeks.

SUMMARY:
This study aims to examine the effect of dramatic play-based activities on bullying behaviors in preschool children; and to evaluate the effects of these activities on empathy levels and social interaction skills, thereby revealing the moderating role of individual and environmental factors in this relationship.

The hypothesis of the research is as follows. H1: Dramatic play has an effect on bullying behaviors in preschool children.

DETAILED DESCRIPTION:
The research will be conducted with all students (3-6 years old) attending a kindergarten affiliated with the Bitlis Provincial Directorate who meet the inclusion criteria. The study will begin with a video animation presentation for preliminary information; this will be followed by dramatic play-based activities aimed at reducing bullying behaviors and supporting empathy and social interaction skills, implemented over 10 weeks. Data will be collected using the "Introductory Information Form," the "Preschool Peer Bullying Scale (Teacher Form)," and the "Bully and Victim Child Behavior Assessment Form."

ELIGIBILITY:
Inclusion Criteria:

* Being in the 3-6 age group
* No learning difficulties
* No communication problems
* Speaking Turkish
* No chronic illnesses
* Suitable/willing to work in a group

Exclusion Criteria:

* Child receiving a chronic diagnosis
* Child leaving school
* Desire to leave work
* Child not adapting to group work

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2025-10-20 (Actual); Primary Completion 2025-12-29 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Identification Information Form | 1 Week
  The form was prepared based on the researchers' previous experiences and the literature to determine the demographic characteristics of the children who constitute the sample of the study. The form contains a total of 11 items to determine information such as the child's age, gender, parental status, family structure, number of siblings, parental education and father's occupation, and duration of preschool education.
Preschool Peer Bullying Scale Teacher Form | 1 Week
  The scale, prepared by Besnili (2019) to investigate peer bullying behaviors among students, is a 14-item, 5-point Likert scale. This scale is completed by the classroom teacher, considering all students in the class. The draft form, initially prepared with 28 items, was reduced to 14 items as a result of the analyses. Scale development was carried out using exploratory and confirmatory factor analyses. For the Exploratory Factor Analysis, data were collected from 279 preschool teachers. In the exploratory factor analysis, Cronbach's Alpha internal consistency coefficients were calculated as .85 for the physical/relational bullying dimension, .79 for the verbal bullying dimension, and .88 for the entire scale. In the Confirmatory Factor Analysis, the other stage of the scale development study, data were collected from 247 different preschool teachers, and in this analysis, the Cronbach's Alpha internal consistency coefficients were calculated as .83 for the physical/relational bullyin
Bully and Victim Child Behavior Assessment Form | 1 Week
  The scale is a measurement tool developed by Özyürek and Kurnaz (2019) to identify bullying, victimizing, and passive bullying behaviors in children in early childhood, based on teachers' observations of children. The scale consists of 32 items in total, with 3 separate dimensions and 13, 14, and 15 items in each dimension. For each item, the teacher must mark one of the "yes" and "no" options that best suit the child they are observing. Answers are scored as (1) for yes and (0) for no. The scale consists of three sub-dimensions: bullying child behaviors, victimizing child behaviors, and passive bullying child behaviors. The internal consistency coefficients of the scale are 0.86 for bullying child behaviors, 0.88 for victimizing child behaviors, and 0.71 for passive bullying child behaviors (Özyürek and Kurnaz, 2019). The sub-dimensions are expressed in the findings section as Bully Child (BCC), Victim Child (VC), and Passive Bully Child (PCC) Behaviors.

SECONDARY OUTCOMES:
Preschool Peer Bullying Scale Teacher Form | 10 Week
  The scale, prepared by Besnili (2019) to investigate peer bullying behaviors among students, is a 14-item, 5-point Likert scale. This scale is completed by the classroom teacher, considering all students in the class. The draft form, initially prepared with 28 items, was reduced to 14 items as a result of the analyses. Scale development was carried out using exploratory and confirmatory factor analyses. For the Exploratory Factor Analysis, data were collected from 279 preschool teachers. In the exploratory factor analysis, Cronbach's Alpha internal consistency coefficients were calculated as .85 for the physical/relational bullying dimension, .79 for the verbal bullying dimension, and .88 for the entire scale. In the Confirmatory Factor Analysis, the other stage of the scale development study, data were collected from 247 different preschool teachers, and in this analysis, the Cronbach's Alpha internal consistency coefficients were calculated as .83 for the physical/relational bullyin
Bully and Victim Child Behavior Assessment Form | 10 Week
  The scale is a measurement tool developed by Özyürek and Kurnaz (2019) to identify bullying, victimizing, and passive bullying behaviors in children in early childhood, based on teachers' observations of children. The scale consists of 32 items in total, with 3 separate dimensions and 13, 14, and 15 items in each dimension. For each item, the teacher must mark one of the "yes" and "no" options that best suit the child they are observing. Answers are scored as (1) for yes and (0) for no. The scale consists of three sub-dimensions: bullying child behaviors, victimizing child behaviors, and passive bullying child behaviors. The internal consistency coefficients of the scale are 0.86 for bullying child behaviors, 0.88 for victimizing child behaviors, and 0.71 for passive bullying child behaviors (Özyürek and Kurnaz, 2019). The sub-dimensions are expressed in the findings section as Bully Child (BCC), Victim Child (VC), and Passive Bully Child (PCC) Behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Güdücü Tüfekci, Study Director — Ataturk University
Locations (1):
- Atatürk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No